CLINICAL TRIAL: NCT04533581
Title: A Japanese Phase 2 Study of ME-401 in Subjects With Relapsed or Refractory Indolent B-cell Non-Hodgkin's Lymphoma (NHL)
Brief Title: Study of ME-401 in Subjects With Relapsed or Refractory Indolent B-cell Non-Hodgkin's Lymphoma (NHL)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ME-401-K02
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Indolent B-cell Non-Hodgkin's Lymphoma
MeSH Terms: interventions — ME-401

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ME-401 (Experimental)
  Interventions: Drug: ME-401

INTERVENTIONS:
Drug: ME-401 — In the first 2 cycles (1 cycle is 28 days), subjects will be administered 60 mg of ME-401 orally once a day on a continuous schedule (CS). After that, subjects will be administered 60 mg of ME-401 orally once a day for the first 7 days, followed by rest for 21 days on an intermittent schedule (IS).

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and pharmacokinetics of ME-401 in the treatment of Japanese participants with Relapsed or Refractory indolent B-Cell Non-Hodgkin's Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 years or older at the submission of the written informed consent form
* Patients that have undergone therapy after at least 2 prior systemic therapies (anti-CD20 Ab, chemo, and so on) for relapsed or refractory B-cell NHL
* Patients who have not undergone phosphatidylinositol 3-kinase (PI3K) inhibitors to date
* Patients who have not undergone Bruton's tyrosine kinase (BTK) inhibitors to date
* Patients with Eastern Cooperative Oncology Group Performance status (ECOG PS) "0 or 1"

Exclusion Criteria:

* Patients with relapsed or refractory B-cell NHL who is categorized into Small lymphocytic lymphoma (SLL), Waldenström's macroglobulinemia (WM), Lymphoplasmacytic lymphoma (LPL) by WHO classification
* Patients who have been histologically confirmed FL Grade 3b transformation from Follicular lymphoma (FL) to an aggressive lymphoma at least once
* Patients with lymphomatous involvement of the central nervous system
* Patients with uncontrolled clinically significant illness
* Patients with active interstitial lung disease or a history thereof

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 2 years
  ORR is measured as the proportion of subjects achieving the best response rating of complete response (CR) or partial response (PR) prior to first progressive disease (PD).

SECONDARY OUTCOMES:
Efficacy of ME-401 as assessed by the duration of response (DOR) | Up to approximately 4 years
Efficacy of ME-401 as assessed by the progression-free survival (PFS) | Up to approximately 4 years
Efficacy of ME-401 as assessed by CR | Up to approximately 4 years
Efficacy of ME-401 as assessed by the Time to treatment failure (TTF) | Up to approximately 4 years
Efficacy of ME-401 as assessed by the objective response rate (ORR) | Up to approximately 4 years
Safety of ME-401 as assessed by the number of participants with treatment-emergent adverse events (TEAEs) | Up to approximately 4 years
Safety of ME-401 as assessed by the time to occurrence of adverse event of special interest (AESI) | Up to approximately 4 years
Plasma concentration level of ME-401 | Up to approximately 4 years

CONTACTS AND LOCATIONS:
Locations (30):
- Japan (30):
  - Anjo Kosei Hospital, Anjo, Aichi-ken
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Japanese Red Cross Nagoya Daini Hospital, Nagoya, Aichi-ken
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Kameda Medical Center, Kamogawa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Gunma University Hospital, Maebashi, Gunma
  - Chugoku Central Hospital, Fukuyama, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Mie University Hospital, Tsu, Mie-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Kindai University Hospital, Sayama, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Tokyo Metropolitan Komagome Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital Of JFCR, Koto-ku, Tokyo
  - Tottori University Hospital, Yonago, Tottori
  - Akita University Hospital, Akita
  - Aomori Prefectural Central Hospital, Aomori
  - Chiba Cancer Center, Chiba
  - Kyushu University Hospital, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Kagoshima University Hospital, Kagoshima
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Japanese Red Cross Kyoto Daini Hospital, Kyoto
  - Okayama University Hospital, Okayama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munakata W, Kumode T, Goto H, Fukuhara N, Shimoyama T, Takeuchi M, Kawakita T, Kubo K, Sawa M, Uchida T, Mishima Y, Ichii M, Hanaya M, Matsumoto A, Kuriki M, Seike T, Izutsu K, Ishizawa K. A phase II study of zandelisib in patients with relapsed or refractory indolent non-Hodgkin lymphoma: ME-401-K02 study. Br J Haematol. 2025 Feb;206(2):541-550. doi: 10.1111/bjh.19994. Epub 2025 Jan 8. PMID 39778876